CLINICAL TRIAL: NCT02067949
Title: The Clinical Outcome and the Cost-effectiveness Analysis of Simvastatin Plus Standard Therapy Versus Standard Therapy Alone in Critically Ill Septic Patient"
Brief Title: Clinical and Economic Outcome of Simvastatin in Critically Ill Septic Patient
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: sara mostafa amin eladawy (Other)
Responsible Party: Sponsor-Investigator, sara mostafa amin eladawy, teaching assistant, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1/2014
Record Dates: First submitted 2014-02-19; First posted 2014-02-20 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- broad spectrum AB +fluids (No Intervention): Control group :50 patients will be treated according to SURVIVING SEPSIS CAMPAIGN BUNDLES
- simvastatin (Active Comparator): 50 patients will be treated according SSCG plus simvastatin as single oral tablet 40 mg / day begin with inclusion in the study and continue until hospital discharge .If the patient is able to swallow; the tablet will be given orally. Otherwise, it will be crushed, suspended in water and administered via any existing enteral feeding or gastric drainage tube. (White R, Bradnam V, 2013)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — single oral tablet 40 mg / day If the patient is able to swallow; the tablet will be given orally. Otherwise, it will be crushed, suspended in water and administered via any existing enteral feeding or gastric drainage tube
  Other Names: Zocor 40 mg
  Arms: simvastatin

SUMMARY:
determination of the effectiveness and the cost-effectiveness of simvastatin(Zocor 40 mg) plus standard therapy (SSCG)versus standard therapy alone in critically ill septic patient from the societal perspective over one year.

DETAILED DESCRIPTION:
Prospective double blinded randomized controlled study Will be carried out at Ain-Shams university hospital Method: - After approval of the research ethics committee of Ain shams University and obtaining consent from each patient, 100 patients newly admitted to the intensive care unit (ICU) diagnosed to have sepsis/severe sepsis defined by American College of Chest Physicians (ACP) *will be randomized by the clinical pharmacist using a computer-generated randomization sequence with a block size of four into two groups.

Group I (Control group):-50 patients will be treated according to "Surviving Sepsis Campaign guidelines (SSCG) (Dellinger, et al. 2013) Group II (Intervention group):-50 patients will be treated according SSCG plus simvastatin.

Outcomes:- Primary outcome measures: 28 day ICU and hospital mortality.

Secondary Outcome Measures:

* Requirement and length of renal replacement therapy, vasoactive agent support or mechanical ventilation
* Total ICU length of stay.(LOS)
* Number of patients alive 3, 6, and 12 months
* Incremental cost effectiveness ratio

ELIGIBILITY:
Inclusion criteria:-

1. Age >18 and less than 70
2. Sepsis for less than 24 hours from ICU admission

Exclusion criteria:-

1. Elderly (defined as older than 70).
2. Pediatrics (defined as younger than 18).
3. Pregnancy and nursing.
4. Unable to receive enteral medications.
5. History of hypersensitivity to the trial drug.
6. Are receiving drugs known to interact with simvastatin.
7. Acute liver failure and chronic liver disease (Child C).
8. High risk of rhabdomyolysis (multiple traumas, crush injuries, extensive burns(>60%), baseline creatinine kinase (CK) ≥ten-times upper limit of normal.
9. Patients with dyslipidemia or Prior statin user.
10. Sever renal impairment (defined as need for replacement therapy )and uncontrolled hypothyroidism
11. Have a history of known or suspected porphyria
12. Are unlikely to survive more than 24 hours

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
28 day ICU and hospital mortality | one year

SECONDARY OUTCOMES:
Number of patients alive 3, 6, and 12 months and incremental cost effectiveness ratio | one year

OTHER OUTCOMES:
ICU hazards | one year
  * Requirement and length of renal replacement therapy, vasoactive agent support or mechanical ventilation
  * Total ICU length of stay.(LOS)

CONTACTS AND LOCATIONS:
Overall Officials: sara M amin, MSC, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university hospital and cairo university hospital, Cairo, Cairo Governorate, Egypt